CLINICAL TRIAL: NCT05286970
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Characteristics of Single Dose Subcutaneous Administration of AK115 in Healthy Subjects
Brief Title: A Clinical Study of AK115 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK115-101
Record Dates: First submitted 2022-03-03; First posted 2022-03-18 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 0.5mg AK115 SC (Experimental): single-dose
  Interventions: Drug: AK115
- 1mg AK115or placebo SC (Experimental): single-dose
  Interventions: Drug: AK115; Drug: Placebo
- 3mg AK115or placebo SC (Experimental): single-dose
  Interventions: Drug: AK115; Drug: Placebo
- 10mg AK115or placebo SC (Experimental): single-dose
  Interventions: Drug: AK115; Drug: Placebo
- 30mg AK115or placebo SC (Experimental): single-dose
  Interventions: Drug: AK115; Drug: Placebo
- 60mg AK115or placebo SC (Experimental): single-dose
  Interventions: Drug: AK115; Drug: Placebo

INTERVENTIONS:
Drug: AK115 — Abdominal subcutaneous injection
Drug: Placebo — Abdominal subcutaneous injection
  Arms: 10mg AK115or placebo SC; 1mg AK115or placebo SC; 30mg AK115or placebo SC; 3mg AK115or placebo SC; 60mg AK115or placebo SC

SUMMARY:
This trial is a randomized, double-blind, placebo-controlled dose escalation phase I trial following single dose subcutaneous administration of AK115 injection.

It aims to evaluate the safety, pharmacokinetic characteristics, pharmacodynamic effect and immunogenicity of single dose of AK115 injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects fully understand the purpose, content, process and possible adverse reactions of the trial, voluntarily participate in the trial, and sign the informed consent before any test procedure;
2. Healthy male and female subjects aged 18-55 years (including 18 and 55 years);
3. Male weight ≥ 50.0kg, female weight ≥ 45.0kg; Body mass index (BMI) = body weight (kg) / height 2 (M2), in the range of 19.0 ~ 26.0kg/m2 (including the critical value);
4. The blood pregnancy test results of female subjects of chidbearing potential during the screening period were negative. During the whole trial period and within 84 days after receiving the inveatigational drug, the subjects and their partners voluntarily take effective contraceptive measures specified in the protocol. Female subjects without childbearing potential need to meet the standards specified in the protocol,
5. The subjects can communicate well with the researchers, understand and comply with the requirements of this trial protocol.

Exclusion Criteria:

1. Allergic to AK115 component and any monoclonal antibody, or have a history of allergies of 3 or more kinds food or drugs ;
2. There are accompanying diseases , or previous serious and chronic diseases and those who have not been cured;
3. The results of physical examination, laboratory examination or ECG examination in the screening period are judged by the researcher to be abnormal and clinically significant;
4. Have a history of transplantation of important organs;
5. Abnormal liver and kidney functions and blood routine, refer to the protocol
6. Hepatitis B surface antigen, hepatitis C antibody, HIV antigen antibody, Treponema pallidum antibody positive;
7. History of alcohol abuse or Drug abusers within 12 months before screening or those with positive urine drug screening results during screening;
8. Blood donation or massive blood loss (> 400ml) or Smoking more than 5 cigarettes per day within 3 months before check-in;
9. Female subjects are in pregnancy or lactation;
10. Use of medications including over-the-counter medication within 14 days before the investigational drug;
11. Participated in the clinical trial of any trial drug within 3 months before the investigational drug or still within 5 half lives of other trial drugs (whichever is longer);
12. Subjects who received monoclonal antibodies or other biological agents within 3 months before investigational drug;
13. Subjects who had received systemic corticosteroids 12 months before screening;
14. Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Incidence and severity classification of adverse events | 0-12week
  Incidence and severity classification of adverse events

SECONDARY OUTCOMES:
Pharmacokinetic parameters of AK115 in healthy subjects | 0-12week
  Pharmacokinetic parameters of AK115 in healthy subjects: peak concentration (Cmax)
Pharmacokinetic parameters of AK115 in healthy subjects | 0-12week
  Pharmacokinetic parameters of AK115 in healthy subjects: time to peak (Tmax)
Pharmacokinetic parameters of AK115 in healthy subjects | 0-12week
  Pharmacokinetic parameters of AK115 in healthy subjects: apparent terminal elimination rate constant（ λ z)
Pharmacokinetic parameters of AK115 in healthy subjects | 0-12week
  Pharmacokinetic parameters of AK115 in healthy subjects: Area under drug time curve (AUC)
Pharmacokinetic parameters of AK115 in healthy subjects | 0-12week
  Pharmacokinetic parameters of AK115 in healthy subjects: apparent total body clearance (CL / F)
Pharmacokinetic parameters of AK115 in healthy subjects | 0-12week
  Pharmacokinetic parameters of AK115 in healthy subjects: apparent distribution volume (VZ / F)
Pharmacokinetic parameters of AK115 in healthy subjects | 0-12week
  Pharmacokinetic parameters of AK115 in healthy subjects: elimination half-life (T1 / 2)
Pharmacokinetic parameters of AK115 in healthy subjects | 0-12week
  Pharmacokinetic parameters of AK115 in healthy subjects: mean residence time (MRT), etc
Changes in serum total nerve growth factor (NGF) levels from baseline. | 0-12 week
  Changes in serum total nerve growth factor (NGF) levels from baseline.
Immunogenicity characteristics: the number and percentage of anti AK115 antibody (ADA) | 0-12week
  Immunogenicity characteristics: the number and percentage of anti AK115 antibody (ADA)
Immunogenicity characteristics: the number and percentage of neutralizing antibody (NAB) positive subjects | 0-12week
  Immunogenicity characteristics: the number and percentage of neutralizing antibody (NAB) positive subjects
Immunogenicity characteristics: time to ADA positive | 0-12week
  Immunogenicity characteristics: time to ADA positive

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan Provincial Hospital of Traditional Chinese Medicine, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Fan YX, Huang Y, Guan R, Li R, Long S, Yang M, Yu B, Wang GQ, Chen P, Gong X, Li B, Xia M, He J. The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Subcutaneous Administration of a Novel Anti-NGF Monoclonal Antibody (AK115) in Healthy Participants: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Phase I Clinical Trial. Drug Des Devel Ther. 2025 Apr 24;19:3225-3235. doi: 10.2147/DDDT.S500902. eCollection 2025. PMID 40297315